CLINICAL TRIAL: NCT05964361
Title: First-in-human Interleukin-15-transpresenting Wilms' Tumor Protein 1-targeting Autologous Dendritic Cell Vaccination in Cancer Patients
Acronym: IL15-TransDC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other); Stichting tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG19-001
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer; Pancreas Cancer; Ovarian Cancer; Liver Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: IL15-transpresenting WT1-targeted Dendritic Cell Vaccine — IL15/IL15Ra/WT1 DC vaccines (8-10 x 10^6 cells in 500 μL saline solution with 5% human albumin) will be administered through intradermal injection at 5 sites (100 μL/site) in the ventromedial region of the upper arm (5-10 cm from the axillary lymph nodes). Injection sites will alternate between left and right arms. WT1/DC vaccines are administered every 2 weeks (+- 3 days) for a total of 6 administrations.
  Other Names: IL15/IL15Ra/WT1 DC vaccine; IL15-transpresenting WT1-targeting DC vaccine

SUMMARY:
The goal of this clinical trial is to investigate a new type of dendritic cell vaccine in patients with refractory or advanced solid tumors of the esophagus, liver, pancreas and ovaries. The main questions it aims to answer are:

* is it feasible to produce and administer these dendritic cell vaccines?
* is treatment with these dendritic cell vaccines safe?

Participants will first need to undergo a leukapheresis procedure to collect the cellular starting material for the dendritic cell vaccine production. The treatment consists of 6 vaccines, administered at biweekly intervals. Participants will be followed-up until 90 days after the last vaccine.

DETAILED DESCRIPTION:
The investigational medicinal product concerns dendritic cells that were engineered to target the tumor antigen Wilms' Tumor-1 (WT1) and in addition transpresent the cytokine IL15 on their cell surface. By inclusion of the IL15-transpresentation mechanism, the intention is to render the dendritic cell more immunogenic (i.e. they have a higher capacity to stimulate the immune system to recognize and attack WT1-expressing cancer cells).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (i.e. date of study entry (T0))
* Age ≥ 18 years at the time of signing informed consent
* Diagnosis with a histologically or cytologically confirmed solid tumor of the pancreas, esophagus, liver or ovaries that is advanced, recurrent or progressing after at least first-line anti-cancer treatment, or for which no alternative standard therapy is available due to intolerance to or refusal of standard-of-care treatment.
* Adequate hematological blood values following previous anti-cancer treatments, as judged by the Principal Investigator
* All treatment-related toxicities must have resolved to CTCAE grade ≤ 2 or must be stable and well controlled with minimal, local or non-invasive intervention, as judged by the Principal Investigator
* Reasonable life expectancy of at least 3 months, as estimated by the Principal Investigator
* At least 1 measurable or evaluable lesion as defined by the latest version of Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) guidelines
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained at the time of screening:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/µL) without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 0.5 x 109/L (500/µL)
  * Platelet count ≥ 100 x 109/L (100,000/µL) without transfusion
  * Hemoglobin ≥ 90 g/L (9 g/dL) (Patients may be transfused to meet this criterion)
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions:

    * Patients with documented liver metastases: AST and ALT ≤ 5 x ULN
    * Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
  * Total bilirubin ≤ 2 x ULN with the following exception:

    * Patients with known Gilbert disease: total bilirubin ≤ 3 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin ≥ 25 g/L (2.5 g/dL)
  * Phosphorus ≥ 0.78 mmol/L
* World Health Organization (WHO) performance status 0-2
* Willing or able to comply with the protocol, as judged by the Principal Investigator
* Women of child bearing potential must have a negative serum or urine pregnancy test at the time of screening. Women of child bearing potential and men must agree to use effective contraception before, during and for at least hundred days after the last study treatment administration.

Exclusion Criteria:

* Use of any investigational agent within 4 weeks before the planned day of leukapheresis
* Corticosteroid treatment within 1 week before leukapheresis, unless the Principal Investigator rationalizes otherwise
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Non-treated brain or meningeal mestases, or priorly treated brain or meningeal metastases with magnetic resonance imaging (MRI) evidence of progression in the last 8 weeks
* Pregnant or breastfeeding. Female subjects who are breastfeeding should discontinue nursing prior to the first dose of study treatment and until at least hundred days after the last study treatment administration
* Any other condition, either physical or psychological, or reasonable suspicion thereof on clinical or special investigation, which contraindicates the use of the vaccine, or may negatively affect patient compliance, or may place the patient at higher risk of potential treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Feasibilty of leukapheresis | Upon completion of leukapheresis, on average 4 weeks after inclusion (baseline)
  Proportion of patients in the intention-to-treat population that had a successful leukapheresis.
Feasibility of IL15/IL15Ra/WT1 DC vaccine production | Upon completion of vaccine production and quality testing (i.e. from leukapheresis until 4 weeks after), on average 8 weeks after inclusion (baseline)
  Proportion of patients in the intention-to-treat population that had successful vaccine production (i.e. production of at least 6 IL-15-transpresenting WT1-targeting DC vaccines meeting all quality control measurements).
Feasibility of study treatment scheme | Study treatment scheme (i.e. from administration of first to 6th vaccine (+- 10 weeks))
  Proportion of patients in the intention-to-treat population who complete the study treatment schedule of 6 IL-15-transpresenting WT1-targeting DC vaccines.
Feasibility of DC vaccine administration (administration of 1st vaccine) | At administration of first vaccine
  Proportion of efficacy evaluable patients (i.e. having received at least 1 vaccine + no major protocol violation) in the intention-to-treat population.
Safety of IL15/IL15Ra/WT1 DC vaccine administration: Related (Severe) Adverse Events ((S)AEs) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  Proportion of patients of the safety population that experienced (S)AEs possibly, probably or definitely related to IL15/IL15Ra/WT1 DC vaccination
Safety of IL15/IL15Ra/WT1 DC vaccine administration: total (S)AEs (number) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  Number of (S)AEs in the safety population (i.e. having received at least 1 DC vaccine)
Safety of IL15/IL15Ra/WT1 DC vaccine administration: total (S)AEs (grade) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  Grade of (S)AEs in the safety population

SECONDARY OUTCOMES:
Indicators of clinical efficacy: Best Overall Response (BOR) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  BOR will be determined per patient as the best response designation during IL-15-transpresenting WT1-targeting DC vaccination, according to the latest version of iRECIST. The response categories are: immune complete response (iCR), immune partial response (iPR), immune stable disease (iSD) and confirmed immune progressive disease (iCPD).
Indicators of clinical efficacy: Duration of Response (DOR) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  DOR will be determined per patient as the time between the date of the first documented tumor response (iPR or iCR) and the subsequent date of the objectively documented disease progression (i.e. date of immune unconfirmed progressive disease (iUPD)) providing that iCPD is confirmed at the next assessment), or death, whichever occurs first. If iUPD occurs, but is disregarded because of later iSD, iPR or iCR, that iUPD date should not be used as the progression event date. At the time of analysis, patients without a recorded event will be censored at the time of the last objective disease assessment.
Indicators of clinical efficacy: Objective Response Rate (ORR) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  ORR is defined as the proportion of patients whose confirmed BOR is either iCR or iPR, where the denominator is the total number of patients in the efficacy evaluable population.
Indicators of clinical efficacy: Disease Control Rate (DCR) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  Proportion of patients with iCR, iPR or iSD, where the denominator is the total number of patients in the efficacy evaluable population.
Indicators of clinical efficacy: Progression-free Survival (PFS) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months. PFS may be updated after study completion.
  PFS will be determined per patient as the time (in months) between the date of diagnosis/study entry and the first date that progression criteria are met (i.e. date of iUPD, providing that iCPD is confirmed at the next assessment). If iUPD occurs, but is disregarded because of later iSD, iPR or iCR, that iUPD date should not be used as the progression event date. At the time of analysis, patients without a recorded event will be censored at the time of the last objective disease assessment.
  If progression is not confirmed and there is no subsequent iSD, iPR or iCR then the iUPD date should still be used in the following scenarios:
  * if the patient stops study treatment because he/she was not considered to be clinically stable or no further response assessments are done (patient refusal or protocol non-compliance or patient death),
  * the next disease assessments are all iUPD and iCPD never occurs.
Indicators of clinical efficacy: Overall Survival (OS) | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months. OS may be updated after study completion.
  OS will be determined per patient as the time (in months) between diagnosis/study entry and death due to any cause. At the time of analysis, patients without a recorded event will be censored at the time they were last known to be alive.
Immunogenicity of vaccination with IL15/IL15Ra/WT1 DC: occurrence of WT1-specfic CD8+ T cells | done on the day of administration of the first vaccine, the fourth vaccine, and on the day at the first follow-up visit following administration of V6 (i.e. +- 10 weeks after V6).
  Occurrence of WT1-specific CD8+ T cells as assessed by TCR sequencing
Evaluation of changes in quality of life: How patients experience the study therapy | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  QLQ-30
Evaluation of changes in quality of life: How patient-reported disease-related symptoms evolve over time | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  QLQ-30
Evaluation of changes in quality of life: How patient-reported quality of life evolves over time | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  QLQ-30
Evaluation of changes in quality of life: How patient-reported quality of life evolves over time | over the entire study duration (i.e. from inclusion (baseline) to end of follow-up, which lasts until 90 days after the last DC vaccine), on average 7 months
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Timon Vandamme, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van den Bergh JM, Lion E, Van Tendeloo VF, Smits EL. IL-15 receptor alpha as the magic wand to boost the success of IL-15 antitumor therapies: The upswing of IL-15 transpresentation. Pharmacol Ther. 2017 Feb;170:73-79. doi: 10.1016/j.pharmthera.2016.10.012. Epub 2016 Oct 21. PMID 27777088
- [Background] Van den Bergh J, Willemen Y, Lion E, Van Acker H, De Reu H, Anguille S, Goossens H, Berneman Z, Van Tendeloo V, Smits E. Transpresentation of interleukin-15 by IL-15/IL-15Ralpha mRNA-engineered human dendritic cells boosts antitumoral natural killer cell activity. Oncotarget. 2015 Dec 29;6(42):44123-33. doi: 10.18632/oncotarget.6536. PMID 26675759